CLINICAL TRIAL: NCT01697072
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo Controlled Study of Rilotumumab (AMG102) With Epirubicin, Cisplatin, and Capecitabine (ECX) as First-line Therapy in Advanced MET-Positive Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: First-Line Treatment for Locally Advanced or Metastatic Mesenchymal Epithelial Transition Factor (MET) - Positive Gastric, Lower Esophageal, or Gastroesophageal Junction (GEJ) Adenocarcinoma
Acronym: RILOMET-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: All Amgen sponsored AMG102 clinical studies were terminated following a pre-planned Data Monitoring Committee safety review of study 20070622.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20070622; 2011-004923-11 (EudraCT Number)
Record Dates: First submitted 2012-09-26; First posted 2012-10-02 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; First Line Treatment Gastroesophageal Junction (GEJ); Gastroesophageal Junction Cancer (GEJ); GEJ Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — rilotumumab; Epirubicin; Cisplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rilotumumab (Experimental): Rilotumumab (15 mg/kg, IV every 21 days) plus Epirubicin, Cisplatin and Capecitabine (ECX)
  Interventions: Drug: Rilotumumab; Drug: Epirubicin; Drug: Cisplatin; Drug: Capecitabine
- Placebo (Placebo Comparator): Rilotumumab-placebo (15 mg/kg, IV every 21 days) plus Epirubicin, Cisplatin and Capecitabine (ECX)
  Interventions: Other: Placebo; Drug: Epirubicin; Drug: Cisplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Rilotumumab — Rilotumumab is a fully human monoclonal antibody immunoglobulin G, type 2 (IgG2) against human hepatocyte growth factor/scatter factor (HGF/SF) that blocks binding of HGF/SF to its receptor MET, inhibiting HGF/MET-driven activities in cells.
  Other Names: AMG102
  Arms: Rilotumumab
Other: Placebo — Placebo
  Other Names: sterile protein-free solution
  Arms: Placebo
Drug: Epirubicin — Epirubicin is an anthracycline cytotoxic agent.
  Other Names: Ellence; Pharmorubicin PFS; Pharmorubicin RDF
Drug: Cisplatin — Cisplatin is a non-cell cycle specific chemotherapeutic agent.
  Other Names: Platinol; Platinol-AQ
Drug: Capecitabine — Capecitabine is an oral fluoropyrimidine.
  Other Names: Xeloda

SUMMARY:
This is a phase 3, multicenter, randomized, double-blind, placebo controlled study of epirubicin, cisplatin & capecitabine (ECX) with rilotumumab or placebo for untreated advanced MET-positive gastric or gastroesophageal junction (GEJ) adenocarcinoma

ELIGIBILITY:
Key Inclusion Criteria:

* Pathologically confirmed unresectable locally advanced or metastatic gastric or GEJ adenocarcinoma •Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1)
* Tumor MET-positive by immunohistochemistry (IHC)
* Evaluable (measurable or non-measurable) disease by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria

Key exclusion criteria:

* Human Epidermal Growth Factor Receptor 2 (HER2) -overexpressing locally advanced or metastatic gastric or GEJ adenocarcinoma •Previous systemic therapy for locally advanced or metastatic gastric or GEJ adenocarcinoma
* Less than 6 months have elapsed from completion of prior neoadjuvant or adjuvant chemotherapy or chemoradiotherapy to randomization
* Previous treatment with anthracyclines must not exceed total cumulative dose of epirubicin of 400 mg/m2
* Squamous cell histology
* Left ventricular ejection fraction (LVEF) < 50%

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years
  To determine if the treatment of rilotumumab in combination with ECX significantly improves overall survival in subjects with unresectable locally advanced or metastatic MET positive gastric or GEJ cancer

SECONDARY OUTCOMES:
PFS | 3 years
  Progression Free Survival (PFS)
TTP | 3 years
  Time to Progression (TTP)
ORR | 3 years
  Objective Response Rate (ORR)
DCR | 3 years
  Disease Control Rate (DCR)
TTR | 3 years
  Time to Response (TTR)
Safety | 3 years
Immunogenicity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (174):
- United States (16):
  - Research Site, Tucson, Arizona
  - Research Site, Aurora, Colorado
  - Research Site, Pueblo, Colorado
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Woodbury, Minnesota
  - Research Site, Henderson, Nevada
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Bedford, Texas
  - Research Site, Dallas, Texas
  - Research Site, Seattle, Washington
- Australia (8):
  - Research Site, Randwick, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Tweed Heads, New South Wales
  - Research Site, Douglas, Queensland
  - Research Site, Elizabeth Vale, South Australia
  - Research Site, Kurralta Park, South Australia
  - Research Site, Heidelberg, Victoria
  - Research Site, Ringwood East, Victoria
- Austria (5):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Liège
  - Research Site, Roeselare
- Brazil (4):
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Pelotas, Rio Grande do Sul
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
- Bulgaria (4):
  - Research Site, Plovdiv
  - Research Site, Shumen
  - Research Site, Sofia
  - Research Site, Varna
- Canada (6):
  - Research Site, Vancouver, British Columbia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
- Czechia (5):
  - Research Site, Hořovice
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Århus C
  - Research Site, Copenhagen
  - Research Site, Odense
- France (13):
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Périgueux
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
- Germany (11):
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Leipzig
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Oldenburg
  - Research Site, Schweinfurt
- Greece (6):
  - Research Site, Athens
  - Research Site, Heraklion - Crete
  - Research Site, Larissa
  - Research Site, Nea Kifissia, Athens
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Nyíregyháza
  - Research Site, Szeged
  - Research Site, Szolnok
- Italy (7):
  - Research Site, Aviano PN
  - Research Site, Brescia
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Roma
- Mexico (4):
  - Research Site, Distrito Federal, Mexico City
  - Research Site, Mexico City, Mexico City
  - Research Site, Cuernavaca, Morelos
  - Research Site, Toluca, State of Mexico
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Konin
  - Research Site, Lodz
  - Research Site, Warsaw
- Portugal (6):
  - Research Site, Aveiro
  - Research Site, Guimarães
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Santa Maria da Feira
  - Research Site, Vila Real
- Romania (7):
  - Research Site, Alba Iulia
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Lasi
  - Research Site, Timișoara
- Russia (8):
  - Research Site, Chelyabinsk
  - Research Site, Ivanovo
  - Research Site, Kazan'
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Vladimir
- Slovakia (4):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Poprad
  - Research Site, Trenčín
- South Africa (5):
  - Research Site, Groenkloof, Gauteng
  - Research Site, Cape Town
  - Research Site, Johannesburg
  - Research Site, Kraaifontein
  - Research Site, Pretoria
- Spain (7):
  - Research Site, Barcelona, Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Terrassa, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Madrid, Madrid
  - Research Site, Pamplona, Navarre
  - Research Site, Oviedo, Principality of Asturias
- Sweden (2):
  - Research Site, Eskilstuna
  - Research Site, Stockholm
- Switzerland (3):
  - Research Site, Bellinzona
  - Research Site, Bern
  - Research Site, Chur
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (9):
  - Research Site, Dnipropetrovsk
  - Research Site, Kharkiv
  - Research Site, Kherson
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Mariupol
  - Research Site, Sumy
  - Research Site, Uzhhorod
- United Kingdom (10):
  - Research Site, Belfast
  - Research Site, Edinburgh
  - Research Site, Guildford
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Northwood
  - Research Site, Salisbury
  - Research Site, Sutton

REFERENCES:
- [Derived] Catenacci DVT, Tebbutt NC, Davidenko I, Murad AM, Al-Batran SE, Ilson DH, Tjulandin S, Gotovkin E, Karaszewska B, Bondarenko I, Tejani MA, Udrea AA, Tehfe M, De Vita F, Turkington C, Tang R, Ang A, Zhang Y, Hoang T, Sidhu R, Cunningham D. Rilotumumab plus epirubicin, cisplatin, and capecitabine as first-line therapy in advanced MET-positive gastric or gastro-oesophageal junction cancer (RILOMET-1): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1467-1482. doi: 10.1016/S1470-2045(17)30566-1. Epub 2017 Sep 25. PMID 28958504
- [Derived] Doshi S, Gisleskog PO, Zhang Y, Zhu M, Oliner KS, Loh E, Perez Ruixo JJ. Rilotumumab exposure-response relationship in patients with advanced or metastatic gastric cancer. Clin Cancer Res. 2015 Jun 1;21(11):2453-61. doi: 10.1158/1078-0432.CCR-14-1661. Epub 2015 Feb 24. PMID 25712685
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com